CLINICAL TRIAL: NCT07253441
Title: A Multiple-arm, Phase 1, Open-label Trial to Determine Dose Strength Equivalence and Effect of Food on To-Be-Marketed Centanafadine QD XR Capsules, Bioequivalence Between Clinical and To-Be-Marketed QD XR Capsules and Relative Bioavailability of To-Be-Marketed QD XR Capsules to SR Tablets in Healthy Adults
Brief Title: A Trial to Characterize Differences in Blood Levels of Different Lots of Centanafadine QD XR and to Understand the Effect of Food on Blood Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00157
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Healthy Volunteers
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (14):
- Cohort 1: CTN 1 × 328.8 mg capsule, Then CTN 2 × 164.4 mg capsules (Experimental): Participants first receive a 1 × 328.8 mg CTN capsule, orally, on Day 1. Then, they receive 2 × 164.4 mg CTN capsules, orally, on Day 4.
  Interventions: Drug: CTN XR (TBM)
- Cohort 1: CTN 2 × 164.4 mg capsule, Then CTN 1 × 328.8 mg capsules (Experimental): Participants first receive 2 × 164.4 mg CTN capsules, orally, on Day 1. Then, they receive 1 × 328.8 mg CTN capsule, orally, on Day 4.
  Interventions: Drug: CTN XR (TBM)
- Cohort 2: CTN Fasted State, Then CTN Fed state (Experimental): Participants first receive 1 × 328.8 mg CTN capsules, orally, in the fasted state, on Day 1. Then, they receive 1 × 328.8 mg CTN capsule, orally, in the fed state, on Day 4.
  Interventions: Drug: CTN XR (TBM)
- Cohort 2: CTN Fed state, Then CTN Fasted state (Experimental): Participants first receive 1 × 328.8 mg CTN capsules, orally, in the fed state, on Day 1. Then, they receive 1 × 328.8 mg CTN capsule, orally, in the fasted state, on Day 4.
  Interventions: Drug: CTN XR (TBM)
- Cohort 3: CTN 200 mg SR, Then CTN164.4 mg XR, Then CTN 400 mg SR, Then CTN 328.8 mg XR (Experimental): Participants first receive CTN 200 mg SR, tablets, orally on Day 1 followed by CTN 164.4 mg XR, capsules, orally on Day 4. Participants then receive CTN 400 mg SR, tablets, orally on Day 7, followed by CTN 328.8 mg XR, capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR
- Cohort 3: CTN 164.4 mg XR, Then CTN 200 mg SR, Then CTN 328.8 mg XR, Then CTN 400 mg SR (Experimental): Participants first receive CTN 164.4 mg XR, capsules, orally on Day 1 followed by CTN 200 mg SR, tablets, orally on Day 4. Participants then receive CTN 328.8 mg XR, capsules, orally on Day 7, followed by CTN 400 mg SR, tablets, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR
- Cohort 3: CTN 400 mg SR, Then CTN 328.8 mg XR, Then CTN 200 mg SR, Then CTN 164.4 mg XR (Experimental): Participants first receive CTN 400 mg SR, tablets, orally on Day 1 followed by CTN 328.8 mg XR, capsules, orally on Day 4. Participants then receive CTN 200 mg SR, tablets, orally on Day 7, followed by CTN 164.4 mg XR, capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR
- Cohort 3: CTN 328.8 mg XR, Then CTN 400 mg SR, Then CTN 164.4 mg XR, Then CTN 200 mg SR (Experimental): Participants first receive CTN 328.8 mg XR, capsules, orally on Day 1 followed by CTN 400 mg SR, tablets, orally on Day 4. Participants then receive CTN 164.4 mg XR, capsules, orally on Day 7, followed by CTN 200 mg SR, tablets, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR
- Cohort 4: CTN 164.4mg (Clin), Then CTN 164.4mg (TBM), Then CTN 328.8mg (Clin) Then CTN 328.8mg (TBM) (Experimental): Participants first receive CTN 164.4 mg XR (Clin), capsules, orally on Day 1 followed by CTN 164.4 mg XR (TBM), capsules, orally on Day 4. Participants then receive CTN 328.8 mg XR (Clin), capsules, orally on Day 7, followed by CTN 328.8 mg XR (TBM), capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN XR (Clin)
- Cohort 4: CTN 164.4mg (TBM), Then CTN 164.4mg (Clin), Then CTN 328.8mg (TBM) Then CTN 328.8mg (Clin) (Experimental): Participants first receive CTN 164.4 mg XR (TBM), capsules, orally on Day 1 followed by CTN 164.4 mg XR (Clin), capsules, orally on Day 4. Participants then receive CTN 328.8 mg XR (TBM), capsules, orally on Day 7, followed by CTN 328.8 mg XR (Clin), capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN XR (Clin)
- Cohort 4: CTN 328.8mg (Clin), Then CTN 328.8mg (TBM), Then CTN 164.4mg (Clin),Then CTN 164.4mg (TBM) (Experimental): Participants first receive CTN 328.8 mg XR (Clin), capsules, orally on Day 1 followed by CTN 328.8 mg XR (TBM), capsules, orally on Day 4. Participants then receive CTN 164.4 mg XR (Clin), capsules, orally on Day 7, followed by CTN 164.4 mg XR (TBM), capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN XR (Clin)
- Cohort 4: CTN 328.8mg (TBM), Then CTN 328.8mg (Clin), Then CTN 164.4mg (TBM) Then CTN 164.4mg (Clin) (Experimental): Participants first receive CTN 328.8 mg XR (TBM), capsules, orally on Day 1 followed by CTN 328.8 mg XR (Clin), capsules, orally on Day 4. Participants then receive CTN 164.4 mg XR (TBM), capsules, orally on Day 7, followed by CTN 164.4 mg XR (Clin), capsules, orally on Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN XR (Clin)
- Cohort 5: CTN 328.8 mg XR (TBM), Then CTN 400 mg SR (Experimental): Participants first receive CTN 328.8 mg XR (TBM), capsules, orally, once a day (QD) from Day 1 to Day 5. Then, they receive CTN 400 mg SR, tablets, orally, from Day 6 to Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR
- Cohort 5: CTN 400 mg SR, Then CTN 328.8 mg XR (TBM) (Experimental): Participants first receive CTN 400 mg SR, tablets, orally from Day 1 to Day 5. Then, they will receive CTN 328.8 mg XR (TBM), capsules, orally, QD from Day 6 to Day 10.
  Interventions: Drug: CTN XR (TBM); Drug: CTN SR

INTERVENTIONS:
Drug: CTN XR (TBM) — Oral capsules
  Other Names: EB-1020
Drug: CTN SR — Oral tablets
  Other Names: EB-1020
  Arms: Cohort 3: CTN 164.4 mg XR, Then CTN 200 mg SR, Then CTN 328.8 mg XR, Then CTN 400 mg SR; Cohort 3: CTN 200 mg SR, Then CTN164.4 mg XR, Then CTN 400 mg SR, Then CTN 328.8 mg XR; Cohort 3: CTN 328.8 mg XR, Then CTN 400 mg SR, Then CTN 164.4 mg XR, Then CTN 200 mg SR; Cohort 3: CTN 400 mg SR, Then CTN 328.8 mg XR, Then CTN 200 mg SR, Then CTN 164.4 mg XR; Cohort 5: CTN 328.8 mg XR (TBM), Then CTN 400 mg SR; Cohort 5: CTN 400 mg SR, Then CTN 328.8 mg XR (TBM)
Drug: CTN XR (Clin) — Oral capsules
  Other Names: EB-1020
  Arms: Cohort 4: CTN 164.4mg (Clin), Then CTN 164.4mg (TBM), Then CTN 328.8mg (Clin) Then CTN 328.8mg (TBM); Cohort 4: CTN 164.4mg (TBM), Then CTN 164.4mg (Clin), Then CTN 328.8mg (TBM) Then CTN 328.8mg (Clin); Cohort 4: CTN 328.8mg (Clin), Then CTN 328.8mg (TBM), Then CTN 164.4mg (Clin),Then CTN 164.4mg (TBM); Cohort 4: CTN 328.8mg (TBM), Then CTN 328.8mg (Clin), Then CTN 164.4mg (TBM) Then CTN 164.4mg (Clin)

SUMMARY:
The purpose of this study is to evaluate the dose strength equivalence of to-be-marketed (TBM) centanafadine (CTN) once daily (QD) extended release (XR) when administered as 2 capsules of 164.4 milligrams (mg) or as a single capsule of 328.8 mg, effect of food on the absorption of the TBM CTN QD XR capsule, and relative bioavailability of clinical (Clin) CTN sustained release (SR) tablets to the TBM CTN QD XR capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 19.0 to 32.0 kilograms per square meter (kg/m^2) (inclusive).
2. In good health as determined by:

   * Medical history
   * Physical examination
   * Electrocardiogram (ECG)
   * Serum/urine chemistry, hematology, and serology tests.
3. Ability to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the investigator, to comply with all the requirements of the trial.

Exclusion Criteria:

1. Clinically significant abnormality in past medical history, or at the screening physical examination, that in the investigator's or sponsor's opinion may place the participant at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug. This includes, but is not limited to, history of or concurrent cardiac, hepatic, renal, neurologic, endocrine, gastrointestinal, respiratory, hematologic, and immunologic disease or cholecystectomy.
2. History of drug and/or alcohol abuse within 2 years prior to screening.
3. History of or current hepatitis or AIDS or carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HCV), or HIV antibodies.
4. History of any significant drug allergy or known or suspected hypersensitivity.
5. A positive urine or breath alcohol test and/or urine drug screen for substance of abuse at screening or upon admission to the trial site.
6. Any participant who, in the opinion of the investigator, should not participate in the trial.

Note: Other protocol-specified Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Cohorts 1, 2, 3, and 4: Maximum Plasma Concentration (Cmax) of CTN | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohorts 1, 2, 3, and 4: Area Under the Plasma Concentration-time Curve Calculated From Time 0 to Time t (AUCt) of CTN | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohorts 1, 2, 3, and 4: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity of CTN | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohort 5: Cmax of CTN | Up to Day 11
Cohort 5: Area Under the Plasma Concentration-time Curve During the Dosing Interval at Steady-state of CTN XR | Up to Day 11
Cohort 5: Area Under the Drug Concentration-time Curve From Time Zero Predose to 24 hours Postdose (AUC0-24h) of CTN SR | 24 Hours postdose up to Day 10
Cohort 5: Minimum Plasma Concentration During a Dosing Interval (Cmin) of CTN | Up to Day 11

SECONDARY OUTCOMES:
Cohorts 1, 2, 3, and 4: Percentage (%) Extrapolated AUC of CTN and its Metabolites | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohorts 1, 2, 3, and 4: AUC0-24h of CTN and its Metabolites | Cohorts 1 and 2: 24 Hours Postdose up to Day 4; Cohorts 3 and 4: 24 Hours Postdose up to Day 10
Cohort 1, 2, 3, and 4: Time to Maximum (peak) Plasma Concentration (tmax) of CTN and its Metabolites | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohort 1, 2, 3, and 4: Apparent Clearance (CL/F) of CTN and its Metabolites | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohort 1, 2, 3, and 4: Volume of Distribution (Vz/F) of CTN | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohort 1, 2, 3, and 4: Terminal Phase Elimination Half-Life (t1/2,z) of CTN and its Metabolites | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12
Cohort 5: Tmax of CTN and its Metabolites | Up to Day 11
Cohort 5: CL/F of CTN | Up to Day 11
All Cohorts: Number of Participants With Adverse Events (AEs) | Cohorts 1 and 2: Up to Day 11; Cohorts 3, 4, and 5: Up to Day 17
All Cohorts: Number of Participants With Potentially Clinically Relevant Laboratory Tests | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12; Cohort 5: Up to Day 11
All Cohorts: Number of Participants With Potentially Clinically Relevant Vital Signs | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12; Cohort 5: Up to Day 11
All Cohorts: Number of Participants With Potentially Clinically Relevant 12-Lead Electrocardiogram (ECG) Tests | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12; Cohort 5: Up to Day 11
All Cohorts: Percentage of Participants With Suicidal Ideation or Suicidal Behavior Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Cohorts 1 and 2: Up to Day 6; Cohorts 3 and 4: Up to Day 12; Cohort 5: Up to Day 11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ICON Lenexa, Lenexa, Kansas
  - ICON Salt Lake City, Millcreek, Utah

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com/